CLINICAL TRIAL: NCT03043430
Title: Anxiolysis for Emergency Department Procedures in Pediatric Patients Using Intranasal Ketamine Compared With Intranasal Midazolam: A Randomized Controlled Trial
Brief Title: Intranasal Ketamine for Anxiolysis in Pediatric Emergency Department Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Research manpower shortage
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, EM Residency, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C.2016.021
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Anxiety; Pediatric ALL; Procedural Anxiety
MeSH Terms: conditions — Anxiety Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medication (ketamine versus midazolam) will be drawn up in unmarked syringe and applied to the patient by mucosal atomization device by a nurse not directly involved in the investigation or the patient's care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): Ketamine 100 mg/mL concentration administered in a single 1.0 mg/kg dose with a maximum of 50mg intranasal via mucosal atomization device.
  Interventions: Drug: Ketamine 100 MG/ML
- Midazolam (Active Comparator): Midazolam 5 mg/mL concentration administered in a single administered in a single 0.3 mg/kg dose with a maximum of 5mg intranasal via mucosal atomization device.
  Interventions: Drug: Midazolam 5 MG/ML

INTERVENTIONS:
Drug: Ketamine 100 MG/ML — Administer ketamine via mucosal atomization device
  Arms: Ketamine
Drug: Midazolam 5 MG/ML — Administer midazolam via mucosal atomization device
  Arms: Midazolam

SUMMARY:
Investigators plan to conduct a randomized, double-blinded, controlled study among pediatric patients requiring minor procedures in the Emergency Department setting. Patients will be randomized to one of two arms of intranasal treatments: ketamine 1.0 mg/kg (K) or midazolam 0.3 mg/kg (M). The primary outcome will be change in anxiety using the Modified Yale Preoperative Anxiety Scale (mYPAS).

DETAILED DESCRIPTION:
The intranasal route of drug delivery is commonly used in Emergency Departments (ED) in pediatric patients. Multiple trials have shown the safety of administration of intranasal ketamine, including studies performed in the ED to treat pain in pediatric patients. The use of ketamine for anxiolysis has not been directly studied; however, ketamine has been shown to have anxiolytic effect at low doses as secondary outcomes when studied. Midazolam has been established as an effective medication to provide analgesia and anxiolysis. Investigators plan to conduct a randomized, double-blinded, controlled study in the Emergency Department. Pediatric patients presenting to the ED with the need for minor procedures who meet the inclusion and exclusion criteria will be consented, and if amenable, will be enrolled. Patients will be randomized to one of two arms of intranasal treatments: ketamine 1.0 mg/kg (K) or midazolam 0.3 mg/kg (M). Patients will be tracked for symptom improvement within the Emergency Department. The primary outcome will be change in anxiety from initial measurement to measurement 5 minutes pre-procedure using the Modified Yale Preoperative Anxiety Scale (mYPAS). Secondary outcomes will include sedation level, adverse events, need for additional medications, change in pain rating, patient and/or parent/guardian satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 2 to 12 years who present to the ED
* Requiring intravenous access
* Requiring laceration repairs
* Requiring incision and drainage of abscesses
* Requiring digital nerve blocks
* Requiring radiological imaging
* Requiring bladder catheterization
* Requiring foreign body removal.

Exclusion Criteria:

* Vital sign abnormalities greater than 20% deviation from age-normalized ranges
* Altered mental status/delirium or intoxication
* Patient or patient's parent/guardian are unwilling to participate or provide informed consent
* Any allergy to ketamine or midazolam
* Patient is female with history of menarche
* Presence of chronic oxygen-dependent pulmonary disease, liver cirrhosis, or renal disease requiring dialysis
* Presence of ischemic heart disease, heart failure, or a history of unstable dysrhythmias
* Presence of intracranial mass or vascular lesion.
* Presence of a history of psychosis or hallucinations
* Weight greater than 100kg
* History of increased intracranial pressure/ hypertensive hydrocephalus within the last 3 months
* Non-English speaking/reading parent/guardian and/or patients
* Patient is acutely psychotic
* Provider feels that patient currently or likely will require chemical and/or physical restraints
* History of prolonged QT-interval
* Nasal trauma
* Epistaxis

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Change in mYPAS | Change in score between initial measurement versus 5 minutes pre-procedure
  Modified Yale preoperative anxiety scale

SECONDARY OUTCOMES:
Change in sedation scale | Change in score between initial measurement versus 5 minutes pre procedure, 5 minutes post procedure, and 5 minutes pre-discharge
  University of Michigan sedation scale
Change in pain rating (Wong-Baker Pain Faces Rating Scale) | Change in score between initial measurement versus 5 minutes pre procedure, 5 minutes post procedure, and 5 minutes pre-discharge
  Wong-Baker Pain Faces Rating Scale
Change in anxiety score (Visual analogue scale) | Change in score between initial measurement versus 5 minutes pre procedure, 5 minutes post procedure, and 5 minutes pre-discharge
  Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Pearson, MD, Principal Investigator — Faculty Physician
Locations (1):
- San Antonio Military Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosseini Jahromi SA, Hosseini Valami SM, Adeli N, Yazdi Z. Comparison of the effects of intranasal midazolam versus different doses of intranasal ketamine on reducing preoperative pediatric anxiety: a prospective randomized clinical trial. J Anesth. 2012 Dec;26(6):878-82. doi: 10.1007/s00540-012-1422-6. Epub 2012 Jun 12. PMID 22688444
- [Background] Roelofse JA, Shipton EA, de la Harpe CJ, Blignaut RJ. Intranasal sufentanil/midazolam versus ketamine/midazolam for analgesia/sedation in the pediatric population prior to undergoing multiple dental extractions under general anesthesia: a prospective, double-blind, randomized comparison. Anesth Prog. 2004;51(4):114-21. PMID 15675259
- [Background] Narendra PL, Naphade RW, Nallamilli S, Mohd S. A comparison of intranasal ketamine and intranasal midazolam for pediatric premedication. Anesth Essays Res. 2015 May-Aug;9(2):213-8. doi: 10.4103/0259-1162.154051. PMID 26417129
- [Background] Khatavkar SS, Bakhshi RG. Comparison of nasal Midazolam with Ketamine versus nasal Midazolam as a premedication in children. Saudi J Anaesth. 2014 Jan;8(1):17-21. doi: 10.4103/1658-354X.125904. PMID 24665234